CLINICAL TRIAL: NCT05416944
Title: Effect of Personalized Perioperative Blood Pressure Management on Postoperative Complications and Mortality in High-risk Patients Having Major Abdominal Surgery: a Multicenter Prospective Randomized Controlled Interventional Clinical Trial
Brief Title: Perioperative Personalized Blood Pressure Management: IMPROVE-multi
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Jena University Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZKSJ0147
Record Dates: First submitted 2022-05-16; First posted 2022-06-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-04

CONDITIONS: Blood Pressure; Intraoperative Hypotension; Postoperative Complications; Surgery; Anesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Masking Description: In patients in the routine management group, the treating anesthesiologists will be blinded to data of preoperative automated blood pressure monitoring to avoid performance bias. Participants are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine management (control) group (No Intervention): Routine intraoperative blood pressure management with a lower intervention threshold of 65 mmHg. In contrast to the patients assigned to the personalized management group, the individual mean nighttime MAP assessed using preoperative automated blood pressure monitoring is not taken into account and the treating anesthesiologists are blinded to the data of preoperative automated blood pressure monitoring.
- Personalized management (intervention) group (Experimental): In patients randomized to the personalized management group, intraoperative mean arterial pressure will be maintained at least at the mean nighttime mean arterial pressure (assessed using preoperative automated blood pressure monitoring) with a minimum mean arterial pressure of 65 mmHg, and maximum mean arterial pressure of 110 mmHg. The perioperative trial intervention period starts with the beginning of the induction of general anesthesia and ends two hours after surgery ends.
  Interventions: Other: Personalized blood pressure management

INTERVENTIONS:
Other: Personalized blood pressure management — Personalized blood pressure management: Intraoperative mean arterial pressure will be maintained at least at the mean nighttime mean arterial pressure (assessed using preoperative automated blood pressure monitoring) with a minimum mean arterial pressure of 65 mmHg, and maximum mean arterial pressure of 110 mmHg.
  Arms: Personalized management (intervention) group

SUMMARY:
Rates of major complications and mortality in the first weeks after surgery remain very high: postoperative mortality is still around 2% in central Europe and the United States. Postoperative deaths are a consequence of postoperative complications. Postoperative complications that are most strongly associated with postoperative death include acute kidney injury and acute myocardial injury. To avoid postoperative complications it is thus crucial to identify and address modifiable risk factors for complications. One of these modifiable risk factors may be intraoperative hypotension. Intraoperative hypotension is associated with major postoperative complications including acute kidney injury, acute myocardial injury, and death. It remains unknown which blood pressure value should be targeted in the individual patient during surgery to avoid physiologically important intraoperative hypotension. In current clinical practice, an absolute mean arterial pressure threshold of 65mmHg is used as a lower "one-size-fits-all" intervention threshold. This "population harm threshold" is based on the results of retrospective studies. However, using this population harm threshold for all patients ignores the obvious fact that blood pressure varies considerably among individuals. In contrast to current "one-size-fits-all" perioperative blood pressure management, the investigators propose the concept of personalized perioperative blood pressure management. Specifically, the investigators propose to test the hypothesis that personalized perioperative blood pressure management reduces the incidence of a composite outcome of acute kidney injury, acute myocardial injury, non-fatal cardiac arrest, and death within 7 days after surgery compared to routine blood pressure management in high-risk patients having major abdominal surgery. The investigators will perform preoperative automated blood pressure monitoring for one night to define individual intraoperative blood pressure targets. Automated blood pressure monitoring is the clinical reference method to assess blood pressure profiles. The mission of the trial is to reduce postoperative morbidity and mortality after major surgery. The vision is to achieve this improvement in patient outcome by using the innovative concept of personalized perioperative blood pressure management. This trial is expected to change and improve current clinical practice and will have a direct impact on perioperative blood pressure management guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients ≥45 years scheduled for elective major abdominal surgery under general anesthesia that is expected to last ≥90 minutes AND
* Presence of ≥1 of the following high-risk criteria:

  * exercise tolerance <4 metabolic equivalents as defined by the guidelines of the American College of Cardiology/American Heart Association
  * renal impairment (serum creatinine ≥1.3 mg/dL or estimated glomerular filtration rate <90 mL/min/1.73 m2 within the last 6 months)
  * coronary artery disease (any stage)
  * chronic heart failure (New York Heart Association Functional Classification ≥II)
  * valvular heart disease (moderate or severe)
  * history of stroke
  * peripheral arterial occlusive disease (any stage)
  * chronic obstructive pulmonary disease (any stage) or pulmonary fibrosis (any stage)
  * diabetes mellitus requiring oral hypoglycemic agent or insulin
  * immunodeficiency due to a disease (e.g., HIV, leukemia, multiple myeloma, solid organ cancer) or therapy (e.g., immunosuppressants, chemotherapy, radiation, steroids [above Cushing threshold])
  * liver cirrhosis (any Child-Pugh class)
  * body mass index ≥30 kg/m2
  * current smoking or 15 pack-year history of smoking
  * age ≥65 years
  * expected anesthesia duration >180 minutes
  * B-type natriuretic peptide (BNP) >80 ng/L or N-terminal B-type natriuretic peptide (NT-proBNP) >200 ng/L within the last 6 months

Exclusion Criteria:

* emergency surgery
* surgery: nephrectomy, liver or kidney transplantation
* status post transplantation of kidney, liver, heart, or lung
* sepsis (according to current Sepsis-3 definition)
* American Society of Anesthesiologists physical status classification V or VI
* pregnancy
* patients on renal replacement therapy
* impossibility of preoperative automated blood pressure monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1272 (Actual)
Dates: Start 2023-02-26 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Composite outcome of major postoperative complications | Postoperative Day 7
  Collapsed composite ("any event versus none") of acute kidney injury, acute myocardial injury (including myocardial infarction), non-fatal cardiac arrest, and death within 7 days after surgery

SECONDARY OUTCOMES:
Composite outcome of major postoperative complications | Postoperative Day 3
  Collapsed incidence of acute kidney injury, acute myocardial injury (including myocardial infarction), non-fatal cardiac arrest, and death within 3 days after surgery
Postoperative acute kidney injury | Postoperative Day 3
  Incidence of acute kidney injury within 3 days after surgery
Postoperative acute kidney injury | Postoperative Day 7
  Incidence of acute kidney injury within 7 days after surgery
Postoperative acute myocardial injury (including myocardial infarction) | Postoperative Day 3
  Incidence of acute myocardial injury (including myocardial infarction) within 3 days after surgery
Postoperative acute myocardial injury (including myocardial infarction) | Postoperative Day 7
  Incidence of acute myocardial injury (including myocardial infarction) within 7 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 3
  Incidence of non-fatal cardiac arrest within 3 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 7
  Incidence of non-fatal cardiac arrest within 7 days after surgery
Postoperative death | Postoperative Day 3
  Incidence of death within 3 days after surgery
Postoperative death | Postoperative Day 7
  Incidence of death within 7 days after surgery
Composite outcome of long-term postoperative complications | Postoperative Day 30
  Collapsed incidence of need for renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, and death within 30 days after surgery
Composite outcome of long-term postoperative complications | Postoperative Day 90
  Collapsed incidence of need for renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, and death within 90 days after surgery
Postoperative need for renal replacement therapy | Postoperative Day 30
  Incidence of need for renal replacement therapy within 30 days after surgery
Postoperative need for renal replacement therapy | Postoperative Day 90
  Incidence of need for renal replacement therapy within 90 days after surgery
Postoperative myocardial infarction | Postoperative Day 30
  Incidence of myocardial infarction within 30 days after surgery
Postoperative myocardial infarction | Postoperative Day 90
  Incidence of myocardial infarction within 90 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 30
  Incidence of non-fatal cardiac arrest within 30 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 90
  Incidence of non-fatal cardiac arrest within 90 days after surgery
Postoperative death | Postoperative Day 30
  Incidence of death within 30 days after surgery
Postoperative death | Postoperative Day 90
  Incidence of death within 90 days after surgery
Postoperative infectious complications | Postoperative Day 7
  Collapsed incidence of fever, respiratory infection, neurological infection, urinary system infection, colitis or infection with Clostridium difficile, endometritis, surgical site infection, deep incisional surgical site infection, organ or space surgical site infection, unknown infection with pathogenic organisms in tissue or fluid, and sepsis within 7 days after surgery
Postoperative fever | Postoperative Day 7
  Incidence of fever within 7 days after surgery
Postoperative respiratory infection | Postoperative Day 7
  Incidence of respiratory infection within 7 days after surgery
Postoperative neurological infection | Postoperative Day 7
  Incidence of neurological infection within 7 days after surgery
Postoperative urinary system infection | Postoperative Day 7
  Incidence of urinary system infection within 7 days after surgery
Postoperative colitis or infection with Clostridium difficile | Postoperative Day 7
  Incidence of colitis or infection with Clostridium difficile within 7
Postoperative endometritis | Postoperative Day 7
  Incidence of endometritis within 7 days after surgery
Postoperative surgical site infection | Postoperative Day 7
  Incidence of surgical site infection within 7 days after surgery
Postoperative deep incisional surgical site infection | Postoperative Day 7
  Incidence of deep incisional surgical site infection within 7 days after surgery
Postoperative organ or space surgical site infection | Postoperative Day 7
  Incidence of organ or space surgical site infection within 7 days after surgery
Postoperative unknown infection with pathogenic organisms in tissue or fluid | Postoperative Day 7
  Incidence of unknown infection with pathogenic organisms in tissue or fluid
Postoperative sepsis | Postoperative Day 7
  Incidence of sepsis within 7 days after surgery
Hospital discharge | Postoperative Day 90
  Time-to-event outcome with the event "hospital discharge"
Unplanned hospital re-admission | Postoperative Day 30
  Incidence of unplanned hospital re-admission within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, M.D., Principal Investigator — Department of Anesthesiology, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Saugel B, Meidert AS, Brunkhorst FM, Bischoff R, Esser J, Mattis M, Naue P, Vogel K, Bergholz A, Flick M, Kroker A, Muller DX, Thomsen KK, Vokuhl C, Wegge M, Bratke S, Graessner M, Jungwirth B, Schmid S, Grundmann CD, Wischermann JM, Kellner P, Steinhaus M, Grusser L, Coldewey SM, Zacharowski K, Meybohm P, Habicher M, Zarbock A, Zitzmann A, Letz S, Neumann C, Larmann J, Renne T, Krause L, Vettorazzi E, Zapf A, Carlstedt A, Sessler DI, Kouz K; IMPROVE-multi Trial Group. Individualized Perioperative Blood Pressure Management in Patients Undergoing Major Abdominal Surgery: The IMPROVE-multi Randomized Clinical Trial. JAMA. 2025 Dec 2;334(21):1893-1904. doi: 10.1001/jama.2025.17235. PMID 41076588
- [Derived] Bergholz A, Meidert AS, Flick M, Krause L, Vettorazzi E, Zapf A, Brunkhorst FM, Meybohm P, Zacharowski K, Zarbock A, Sessler DI, Kouz K, Saugel B. Effect of personalized perioperative blood pressure management on postoperative complications and mortality in high-risk patients having major abdominal surgery: protocol for a multicenter randomized trial (IMPROVE-multi). Trials. 2022 Nov 17;23(1):946. doi: 10.1186/s13063-022-06854-0. PMID 36397173